CLINICAL TRIAL: NCT03052127
Title: A Phase 1B/2 Open-Label, Ascending Single and Repeat Dose Clinical Trial Designed to Evaluate the Safety and Efficacy of Light-activated AU-011 for the Treatment of Subjects With Small Primary Choroidal Melanoma
Brief Title: Study in Subjects With Small Primary Choroidal Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AU-011-101
Record Dates: First submitted 2017-02-06; First posted 2017-02-14 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Uveal Melanoma; Ocular Melanoma; Choroidal Melanoma
Keywords: Uveal melanoma; Eye cancer; Ocular melanoma; Choroidal melanoma
MeSH Terms: conditions — Uveal Melanoma; Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (12):
- Single Low Dose Light-activated AU-011 (Experimental): Low dose Light-activated AU-011 followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Single Medium Dose Light-activated AU-011 (Experimental): Medium dose Light-activated AU-011 followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Single High Dose Light-activated AU-011 (Experimental): High dose Light-activated AU-011 followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- 2 Repeat Medium Dose Light-activated AU-011 (Experimental): 2 repeat medium doses of Light-activated AU-011 each followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- 3 Repeat Medium Dose Light-activated AU-011 (Experimental): 3 repeat medium doses of Light-activated AU-011 followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Single High Dose Light-activated AU-011 x 2 lasers (Experimental): High dose Light-activated AU-011 followed by two laser light applications
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- 3 Repeat High Dose Light-activated AU-011 (Experimental): 3 repeat high doses of Light-activated AU-011 each followed by a single laser light application
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- 3 Repeat High Dose Light-activated AU-011 x 2 lasers (Experimental): 3 repeat high doses of Light-activated AU-011 each followed by two laser light applications
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Expansion 3 Repeat High Dose Light-activated AU-011 x 2 lasers (Experimental): Expansion of 3 repeat high doses of Light-activated AU-011 each followed by two laser light applications (up to 12 additional subjects)
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Observation until Documented Growth of Tumor (Experimental): Observation until documented growth of tumor and then treatment with 2 cycles each of 3 repeat high doses of Light-activated AU-011 each followed by two laser light applications
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- 2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 lasers (Experimental): 2 cycles each of 3 repeat high doses of Light-activated AU-011 each followed by two laser light applications
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation
- Exp: 2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers (Experimental): 2 cycles each of 3 repeat high doses of Light-activated AU-011 each followed by two laser light applications in subjects with evidence of documented tumor growth prior to study entry
  Interventions: Drug: Light-activated AU-011; Device: Laser Activation

INTERVENTIONS:
Drug: Light-activated AU-011 — Study treatment
Device: Laser Activation — Study treatment
  Other Names: PDT Laser

SUMMARY:
The primary objective is to assess the safety, immunogenicity and efficacy of one of three dose levels and repeat dose regimens of Light-activated AU-011 and one or two laser applications for the treatment of subjects with primary choroidal melanoma.

DETAILED DESCRIPTION:
This is a phase 1B/2 open-label, ascending single and repeat dose clinical trial designed to evaluate the safety and efficacy of Light-activated AU-011 for the treatment of subjects with small primary choroidal melanoma.

Throughout the study, subjects will be monitored through medical and ophthalmic assessments. Subjects will be followed for a total of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of choroidal melanoma

Exclusion Criteria:

* Have known contraindications or sensitivities to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Narvekar, MBBS, Study Director — Aura Biosciences
Locations (13):
- United States (13):
  - Retina Associates SW, P.C., Tucson, Arizona
  - UCLA Jules Stein Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Retina Consultants of Sacramento, Sacramento, California
  - Colorado Retina Associates, Denver, Colorado
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W. K. Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Associated Retinal Consultants, PC, Royal Oak, Michigan
  - Retina Center, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - Retina Consultants of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 57 participants with Primary Choroidal Melanoma at 15 sites in the USA were enrolled and 56 were treated with at least 1 dose of AU-011 at 3 dose levels and repeat dose regimens in 1 or 2 treatment cycles with 1 or 2 laser applications.
Pre-assignment Details: This open-label, multicenter, dose escalation trial with expansion cohorts was designed to evaluate the safety, immunogenicity, and efficacy of up to 2 treatment cycles of intravitreal (IVT) AU-011 aimed to enroll approximately 60 participants with small primary CM. The tables were created for overall and by cohort as part of the study design. Each study participant contributed only 1 eye (study eye).
Groups:
- Cohort 1 (Light-activated AU-011): Low dose (20 µg) Light-activated AU-011 followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 2 (Single Medium Dose Light-activated AU-011): Medium dose (40 µg) Light-activated AU-011 followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 3 (Single High Dose Light-activated AU-011): High dose (80 µg) Light-activated AU-011 followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 4 (2 Repeat Medium Dose Light-activated AU-011): 2 repeat medium doses (40 µg) of Light-activated AU-011 each followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 5 (3 Repeat Medium Dose Light-activated AU-011): 3 repeat medium doses (40 µg) of Light-activated AU-011 followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers): High dose (80 µg) Light-activated AU-011 followed by two laser light applications
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 7 (3 Repeat High Dose Light-activated AU-011): 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by a single laser light application
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers): 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers): Expansion of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications once for 3 weeks with potential for retreatment
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 10 (Observation Until Documented Growth of Tumor): Expansion - Observation until documented growth of tumor and then treatment with 2 cycles each of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011 x 2 Lasers): Expansion - 2 cycles each of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011 x 2 Lasers): Expansion: 2 cycles each of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications in subjects with evidence of documented tumor growth prior to study entry
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
Period: Overall Study
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011 x 2 Lasers)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13
Completed | 2 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 7 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 5 | 3 | 5 | 13
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Discontinuation by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 5 | 13
Not completed — Inability to comply with trial requirements | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 restrictions and Investigator discretion | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population defined as all enrolled participants, whether or not they received an administration of AU-011 was used for baseline characteristics.
Groups:
- Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers): Expansion - 2 cycles each of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers): Expansion: 2 cycles each of 3 repeat high doses (80 µg) of Light-activated AU-011 each followed by two laser light applications in subjects with evidence of documented tumor growth prior to study entry
  Light-activated AU-011: Study treatment
  Laser Activation: Study treatment
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (6.51) | 61.3 (10.02) | 65.3 (5.13) | 50.3 (9.07) | 52.0 (11.53) | 56.0 (13.11) | 48.0 (14.93) | 57.0 (13.00) | 57.1 (10.47) | 58.0 (9.64) | 68.8 (4.66) | 49.5 (17.85) | 55.7 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 6 | 1 | 3 | 6 | 25
  Male | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 2 | 6 | 2 | 2 | 7 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 12 | 3 | 5 | 13 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13 | 57
Baseline Tumor Characteristics [Mean (Standard Deviation); unit: millimeters] — Tumor thickness assessed using B-scan/ultrasound (reported by independent reading center). Tumor largest basal diameter, distance from fovea, distance from nerve edge - assessed by fundus photography (reported by independent reading center).
  millimeters
    Tumor lesion thickness | 1.9 (0.58) | 2.7 (0.73) | 2.4 (0.35) | 2.0 (0.26) | 2.2 (0.23) | 2.2 (0.15) | 2.2 (0.54) | 2.9 (0.32) | 2.1 (0.42) | 2.6 (0.38) | 1.9 (0.38) | 1.8 (0.6) | 2.1 (0.52)
    Tumor largest basal diameter | 7.7 (2.2) | 8.4 (1.4) | 7.7 (1.4) | 7.8 (1.7) | 8.9 (2.2) | 7.5 (1.2) | 7.9 (1.0) | 12.3 (1.5) | 9.5 (2.7) | 9.7 (2.1) | 7.5 (1.1) | 7.9 (1.5) | 8.6 (2.1)
    Distance from fovea | 4.8 (0.71) | 3.8 (2.4) | 4.6 (0.95) | 4.9 (3.3) | 1.8 (2.1) | 3.8 (1.8) | 5.0 (5.0) | 6.1 (2.9) | 2.9 (2.0) | 3.9 (3.7) | 3.6 (4.4) | 0.9 (0.7) | 3.2 (2.7)
    Distance from nerve edge | 7.7 (1.4) | 2.1 (2.7) | 6.5 (2.7) | 2.2 (3.3) | 1.7 (1.5) | 6.5 (1.4) | 4.0 (5.1) | 4.5 (7.6) | 2.6 (2.2) | 3.0 (1.8) | 3.8 (3.6) | 2.9 (1.5) | 3.6 (3.0)
Baseline Risk factors [Count of Participants; unit: Participants] — Risk factors for diagnosis and growth/progression of primary choroidal melanoma include documented growth, subretinal fluid, presence of orange pigment, decreased vision caused by the tumor, and visual symptoms such as flashes/floaters etc.
  Participants
    Documented Growth | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 7 | 0 | 5 | 13 | 35
    Subretinal fluid | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 11 | 54
    Orange pigmentation | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 10 | 2 | 5 | 8 | 46
    Vision loss | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 6 | 12
    Flashes or floaters | 1 | 2 | 0 | 1 | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 5 | 27
Visual Acuity Scores (ETDRS Letters) in Both Eyes [Mean (Standard Deviation); unit: letters on ETDRS scale] — Visual Acuity assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) method in the intention-to treat (ITT) population
  letters on ETDRS scale
    Study Eye | 89.7 (0.58) | 81.0 (14.18) | 87.3 (4.93) | 88.3 (14.36) | 75.7 (10.69) | 87.0 (3.61) | 87.3 (5.13) | 82.7 (3.21) | 82.9 (10.13) | 86.0 (12.7) | 81.2 (6.34) | 77.9 (11.83) | 82.6 (9.83)
    Fellow Eye | 86.3 (4.62) | 72.7 (17.62) | 80.0 (13.86) | 91.7 (4.73) | 90.3 (1.53) | 86.0 (7.21) | 89.0 (2.65) | 75.0 (19.97) | 88.6 (7.08) | 91.0 (4.58) | 86.2 (7.16) | 85.1 (9.02) | 85.7 (9.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability] of Light-activated AU-011
Description: Adverse events will be summarized by presenting the number and percentage of participants having any adverse event.
Time Frame: Informed consent through 1-2 years
Population: All participants who received at least 1 dose of AU-011 were used for safety analyses.
  Adverse events were defined as events that were new or worsened during the treatment period.
  AEs were coded using the MedDRA Version 20.0 and were graded according to the National Center Institute Common Terminology Criteria for AEs (NCI-CTCAE criteria [v4.03]).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
Participants | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13

2. Secondary Outcome: Immunogenicity (Anti-AU-011 Antibody Analysis)
Description: Percentage of Participants with Anti-AU-011 Antibodies (Anti-Drug Antibody, ADA)
Time Frame: Screening to various time points through 24 months
Population: Subjects who had at least one post-AU-011 dose result were defined in this study as being evaluable for assessment of treatment-induced antibodies to AU-011.
  Negative ADA refers to all negative values at baseline and post-treatment Treatment-induced ADA refers to negative value at baseline and at least 1 positive result post-treatment Treatment-unaffected ADA refers to positive value at baseline and at least 1 reported result post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
Participants
  Negative ADA | 2 | 1 | 3 | 1 | 0 | 2 | 2 | 0 | 4 | 1 | 0 | 1
  Treatment-induced ADA | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 3 | 8 | 1 | 5 | 11
  Treatment-unaffected ADA | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Tumor Size (Thickness) Measured by Ultrasonography [Efficacy]
Description: Change from Baseline in maximum tumor thickness (in millimeters) assessed at each study visit using B-scan ultrasound.
Time Frame: Change from baseline following treatment and at each subsequent visit through Week 52
Population: The intention-to-treat (ITT) population was defined as all enrolled participants, whether or not they received an administration of AU-011.
  Note: The Baseline tumor thickness (TT) values reported for Cohort 10 in the table below (i.e., 2.583 (0.542)) includes only 2 participants who received AU-011. However, the TT values reported in the Baseline Characteristics table (i.e., 2.6 (0.38) includes 3 participants enrolled in the study (ITT population).
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13
millimeters
  Baseline: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Baseline | 1.872 (0.576) | 2.678 (0.734) | 2.389 (0.347) | 2.033 (0.265) | 2.233 (0.233) | 2.233 (0.153) | 2.167 (0.536) | 2.889 (0.320) | 2.072 (0.417) | 2.583 (0.542) | 1.920 (0.384) | 1.826 (0.604)
  Day 2 (Visit 3): number analyzed (Participants) | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2 (Visit 3) | -0.56 (0.069) | 0 (0.100) | -0.011 (0.038) | -0.033 (0) |  |  |  |  |  |  |  |
  Day 8 (Visit 4): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 12 | 2 | 5 | 13
  Day 8 (Visit 4) | -0.042 (0.012) | 0.022 (0.084) | 0.044 (0.084) | 0.044 (0.039) | -0.011 (0.039) | -0.050 (0.071) | 0.067 (0.033) | -0.044 (0.077) | -0.019 (0.73) | 0.017 (0.024) | 0.013 (0.051) | 0.018 (0.059)
  Day 15 (Visit 6): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 12 | 2 | 5 | 13
  Day 15 (Visit 6) | -0.017 (0.024) | 0.044 (0.135) | 0.033 (0.133) | 0.044 (0.019) | 0.033 (0.067) | 0 (0.047) | 0.044 (0.084) | 0.078 (0.051) | -0.028 (0.107) | 0.017 (0.165) | 0.007 (0.159) | 0.021 (0.062)
  Day 29 (Visit 8): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 4 | 13
  Day 29 (Visit 8) | -0.061 (0.151) | 0.056 (0.158) | 0.067 (0.240) | -0.044 (0.184) | 0.011 (0.126) | 0.033 (0.120) | 0.078 (0.164) | 0.111 (0.138) | -0.022 (0.109) | 0 (0.047) | 0.017 (0.104) | 0.018 (0.069)
  Week 8 (Visit 10): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 2 | 5 | 13
  Week 8 (Visit 10) | -0.006 (0.177) | 0.267 (0.200) | 0.111 (0.337) | -0.111 (0.204) | 0.078 (0.039) | 0.056 (0.126) | 0.21 (0.184) | 0.122 (0.126) | -0.012 (0.111) | 0.150 (0.071) | 0.020 (0.119) | -0.010 (0.080)
  Week 12 (Visit 11): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 0 | 5 | 13
  Week 12 (Visit 11) | 0.033 (0.233) | 0.333 (0.285) | 0.144 (0.252) | -0.156 (0.269) | 0.022 (0.077) | -0.100 (0.120) | 0.333 (0.208) | 0.233 (0.219) | 0.028 (0.175) |  | 0.027 (0.130) | -0.049 (0.141)
  Week 26 (Visit 12): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 12
  Week 26 (Visit 12) | -0.117 (0.118) | 1.067 (1.393) | 0.267 (0.635) | -0.044 (0.154) | 0.211 (0.278) | 0.078 (0.250) | 0.733 (0.569) | 0.667 (0.839) | 0.092 (0.25) | 1.20 (1.273) | 0.087 (0.112) | -0.117 (0.400)
  Week 39 (Visit 13): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 1 | 2 | 11 | 2 | 5 | 12
  Week 39 (Visit 13) | -0.067 (0.047) | 0.978 (0.956) | -0.067 (0.094) | -0.333 (0.384) | 0.322 (0.320) | 0.044 (0.217) | 0.133 | 0.300 (0.141) | 0.164 (0.194) | 2.350 (2.616) | 0.147 (0.216) | -0.039 (0.401)
  Week 52 (Visit 14): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 9 | 2 | 5 | 12
  Week 52 (Visit 14) | -0.067 (0.094) | 0.189 (1.151) | -0.067 (0.047) | -0.300 (0.449) | 0.500 (0.404) | 0.156 (0.356) | 0.433 (0.404) | 0.456 (0.320) | 0.222 (0.254) | 2.750 (2.993) | 0.247 (0.315) | 0.128 (0.683)

4. Secondary Outcome: Tumor Size (Diameter) Measured by Fundus Photography [Efficacy]
Description: Change from Baseline in tumor Largest Basal Diameter (LBD) assessed at each study visit based on fundus photos (millimeters) in participants treated with AU-011.
Time Frame: Change from baseline following treatment and at each subsequent visit through Week 52
Population: The intention-to-treat (ITT) population was defined as all enrolled participants, whether or not they received an administration of AU-011.
  Note: The Baseline tumor Largest Basal Diameter (LBD) values reported for Cohort 10 in the table below (i.e., 10.088 (2.825)) includes only 2 participants who received AU-011. However, the LBD values reported in the Baseline Characteristics table (i.e., 9.7 (2.1) includes 3 participants enrolled in Cohort 10 (ITT population).
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13
millimeters
  Baseline: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Baseline | 7.740 (2.197) | 8.350 (1.400) | 7.700 (1.375) | 7.815 (1.681) | 8.853 (2.146) | 7.492 (1.227) | 7.927 (1.030) | 12.257 (1.533) | 9.533 (2.688) | 10.088 (2.825) | 7.502 (1.058) | 7.869 (1.532)
  Day 2 (Visit 3): number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 1 | 12 | 1 | 4 | 11
  Day 2 (Visit 3) | 0.203 (0.414) | 0.280 (0.156) | 0.023 (0.253) | 0.092 (0.226) | -0.308 (0.103) | 0.063 (0.201) | 0.083 (0.131) | 0.410 | -0.161 (0.496) | 0.285 | -0.021 (0.086) | -0.012 (0.234)
  Day 8 (Visit 4): number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 12 | 2 | 5 | 13
  Day 8 (Visit 4) | 0.070 (0.198) | -0.035 (0.347) | 0.225 (0.628) | 0.383 (0.160) | 0.015 (0.566) | 0.080 (0.339) | 0.105 (0.102) | 0.340 (0.149) | -0.154 (0.552) | 0.67 (0.414) | 0.083 (0.215) | 0.168 (0.329)
  Day 9 (Visit 5): number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 0 | 3 | 2 | 11 | 2 | 4 | 11
  Day 9 (Visit 5) |  |  |  | 0.473 (0.464) | -0.007 (0.363) |  | 0.265 (0.141) | 0.918 (0.378) | -0.175 (0.482) | -0.010 (0.481) | 0.060 (0.048) | 0.066 (0.197)
  Day 15 (Visit 6): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 12 | 1 | 3 | 12
  Day 15 (Visit 6) | 0.060 (0.007) | 0.147 (0.140) | 0.417 (0.212) | 0.225 (0.065) | 0.087 (0.253) | 0.500 (0.120) | 0.285 (0.069) | 0.730 (0.644) | -0.130 (0.579) | 0.250 | -0.073 (0.129) | 0.175 (0.319)
  Day 16 (Visit 7): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 10 | 1 | 3 | 11
  Day 16 (Visit 7) |  |  |  |  | -0.010 (0.426) |  | 0.317 (0.025) | 1.120 (1.004) | -0.049 (0.899) | 0.245 | 0.037 (0.928) | 0.265 (0.342)
  Day 29 (Visit 8): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 1 | 8 | 0 | 3 | 9
  Day 29 (Visit 8) | -0.165 (0.184) | 0.003 (0.339) | 0.625 (0.435) | 0.580 (0.180) | 0.198 (0.610) | 0.115 (0.050) | 0.343 (0.060) | 1.660 | 0.019 (0.498) |  | 0.223 (0.335) | 0.199 (0.549)
  Week 6 (Visit 9): number analyzed (Participants) | 0 | 0 | 3 | 3 | 3 | 2 | 2 | 1 | 7 | 0 | 2 | 11
  Week 6 (Visit 9) |  |  | 0.730 (0.265) | 0.627 (0.477) | 0.072 (0.362) | 0.285 (0.021) | 0.333 (0.032) | 0.895 | 0.626 (0.918) |  | -0.222 (0.251) | 0.293 (0.369)
  Week 8 (Visit 10): number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 4 | 1 | 3 | 11
  Week 8 (Visit 10) | -0.472 (0.774) | 0.273 (0.475) | 0.288 (0.239) | 0.807 (0.478) | 0.168 (0.339) | 0.122 (0.214) | 0.970 (0.599) | 2.56 | 0.981 (1.641) | -0.395 | 0.033 (0.287) | 0.314 (0.406)
  Week 12 (Visit 11): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 8 | 2 | 4 | 12
  Week 12 (Visit 11) | -0.468 (0.842) | 0.347 (0.289) | 0.657 (0.144) | 0.963 (0.752) | 0.103 (0.450) | 0.497 (0.138) | 0.930 (0.552) | 1.013 (0.067) | 0.534 (1.173) | -0.115 (0.064) | 0.503 (0.236) | 0.657 (0.703)
  Week 26 (Visit 12): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 10 | 2 | 5 | 11
  Week 26 (Visit 12) | 0.085 (0.212) | -0.032 (0.618) | 0.413 (0.350) | 0.998 (0.959) | 0.412 (1.086) | 0.695 (0.785) | 2.70 (0.961) | 2.857 (1.425) | 1.381 (1.223) | 0.490 (0.212) | 0.738 (0.499) | 0.666 (0.803)
  Week 39 (Visit 13): number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 1 | 8 | 2 | 3 | 8
  Week 39 (Visit 13) | 0.070 (0.332) | 0.805 (0.781) | 0.545 (0.332) | 0.740 (0.014) | 0.445 (0.507) | 0.730 (0.692) | 2.552 (1.552) | 2.635 | 1.342 (1.200) | 0.065 (0.481) | 0.977 (0.365) | 1.224 (0.952)
  Week 52 (Visit 14): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 7 | 1 | 5 | 10
  Week 52 (Visit 14) | 0.230 (0.453) | 0.827 (0.725) | 0.427 (0.180) | 1.605 (1.286) | 0.853 (1.199) | 0.937 (0.814) | 2.993 (1.095) | 1.853 (0.661) | 1.774 (1.254) | 1.630 | 1.197 (0.919) | 1.457 (1.456)

5. Secondary Outcome: Best Corrected Visual Acuity Measured by ETDRS Method [Efficacy] in Study Eye
Description: Change from Baseline in Best Corrected Visual Acuity using ETDRS letters in Study Eye at each study visit.
Time Frame: Change from baseline following treatment and at each subsequent visit through Week 52
Population: The intention-to-treat (ITT) population was defined as all enrolled participants, whether or not they received an administration of AU-011.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011 x 2 Lasers)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 13
ETDRS letters
  Baseline | 89.7 (0.58) | 81.0 (14.18) | 87.3 (4.93) | 88.3 (14.36) | 75.7 (10.69) | 87.0 (3.61) | 87.3 (5.13) | 82.7 (3.21) | 82.9 (10.13) | 86.0 (12.77) | 81.2 (6.34) | 77.9 (11.83)
  Day 2 (Visit 3): number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 11 | 2 | 5 | 13
  Day 2 (Visit 3) | -5.3 (4.04) | -4.0 (12.17) | -14.3 (17.04) | -4.7 (9.07) | -1.0 (1.41) | -11.0 (6.56) | 2.0 (2.00) | -15.0 (16.52) | -4.1 (9.49) | -14.0 (5.66) | -10.2 (16.63) | -0.5 (4.67)
  Day 8 (Visit 4): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Day 8 (Visit 4) | -2.3 (2.52) | 5.3 (3.21) | -3.3 (4.93) | -1.3 (2.08) | -4.3 (4.62) | -6.3 (8.39) | 3.3 (2.52) | -13.0 (23.4) | 0.1 (3.32) | 0.5 (3.54) | 0.4 (3.36) | 1.6 (4.29)
  Day 9 (Visit 5): number analyzed (Participants) | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 3 | 12 | 2 | 5 | 13
  Day 9 (Visit 5) |  |  |  | -3.0 (6.56) | -9.0 (2.83) |  | 0.3 (4.16) | -30.0 (47.76) | -3.4 (8.16) | -0.5 (4.95) | -8.2 (12.50) | -6.2 (13.01)
  Day 15 (Visit 6): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Day 15 (Visit 6) | -2.0 (2.65) | 4.0 (3.61) | -7.0 (8.19) | -6.0 (7.94) | -13.0 (7.00) | -13.3 (17.95) | 0 (8.00) | -4.7 (8.96) | -4.0 (6.97) | 3.5 (2.12) | -20.6 (31.71) | -7.1 (16.32)
  Day 16 (Visit 7): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 3 | 11 | 2 | 5 | 13
  Day 16 (Visit 7) |  |  |  |  | -15.7 (10.26) |  | -1.3 (11.68) | -17.3 (12.06) | -17.0 (16.15) | 0 (2.83) | -28.0 (28.02) | -8.8 (15.24)
  Day 29 (Visit 8): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Day 29 (Visit 8) | -4.3 (5.86) | -0.3 (4.73) | -9.7 (8.33) | -13.7 (7.23) | -9.3 (1.15) | -11.0 (12.12) | -13.7 (23.46) | -10.0 (9.54) | -26.0 (29.60) | -27.5 (7.78) | -26.0 (25.81) | -12.0 (16.38)
  Week 6 (Visit 9): number analyzed (Participants) | 1 | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 2 | 5 | 13
  Week 6 (Visit 9) | -26.0 |  | -2.3 (4.51) | -9.0 (7.55) | -10.0 (7.55) | -9.0 (15.52) | -5.3 (9.5) | -10.0 (10.15) | -8.7 (7.40) | -13.5 (17.68) | -18.6 (23.39) | -7.5 (16.10)
  Week 8 (Visit 10): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Week 8 (Visit 10) | -6.3 (2.08) | 0.3 (3.79) | -7.3 (6.03) | -5.3 (4.93) | -14.7 (14.57) | -11.7 (21.36) | -2.0 (2.65) | -5.3 (2.08) | -6.6 (8.2) | -4.0 (7.07) | -14.2 (23.12) | -8.7 (16.18)
  Week 12 (Visit 11): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 3 | 5 | 12
  Week 12 (Visit 11) | -2.3 (3.79) | 4.0 (1.00) | -3.0 (3.00) | -4.0 (1.73) | -12.0 (13.23) | -11.0 (21.63) | -1.3 (4.04) | -0.7 (3.06) | -3.8 (4.39) | 0 (3.0) | -14.2 (21.32) | -9.4 (15.17)
  Week 26 (Visit 12): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 12 | 2 | 5 | 13
  Week 26 (Visit 12) | 0.3 (3.06) | 0.3 (2.08) | -3.0 (2.65) | -2.7 (1.53) | -1.7 (16.01) | -11.3 (21.39) | -2.0 (6.56) | -0.7 (4.51) | -1.5 (4.36) | 0 (4.24) | -13.0 (18.64) | -9.8 (13.57)
  Week 39 (Visit 13): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 2 | 2 | 11 | 2 | 5 | 12
  Week 39 (Visit 13) | -4.0 (5.66) | -11.0 (20.78) | 0.5 (0.71) | -11.7 (4.73) | -7.0 (23.07) | -9.7 (20.31) | -36.0 (38.18) | -1.0 (0.0) | -8.7 (25.43) | -6.5 (12.02) | -16.8 (19.27) | -10.6 (15.14)
  Week 52 (Visit 14): number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 10 | 2 | 5 | 12
  Week 52 (Visit 14) | -3.0 (2.83) | -18.7 (34.93) | 1.5 (2.12) | -11.3 (4.73) | -7.7 (22.01) | -10.7 (22.85) | -8.3 (13.65) | -1.0 (6.08) | -15.7 (26.56) | -25.0 (11.31) | -17.2 (20.91) | -16.1 (18.34)

ADVERSE EVENTS:
Time Frame: 12 to 24 months
Description: Safety analyses were performed on all participants who received at least 1 dose of AU-011. Only 56 of the 57 enrolled participants received at least 1 dose of AU-011.
  Adverse events (AEs) were defined as events that were new or worsened during the treatment period.
  AEs were coded using the MedDRA Version 20.0 and were graded according to the National Center Institute Common Terminology Criteria for AEs (NCI-CTCAE criteria [v4.03]).
Arm/Group | Cohort 1 (Light-activated AU-011) | Cohort 2 (Single Medium Dose Light-activated AU-011) | Cohort 3 (Single High Dose Light-activated AU-011) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) | Cohort 10 (Observation Until Documented Growth of Tumor) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/12 | 0/2 | 0/5 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/12 | 0/2 | 2/5 | 1/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 12/12 | 2/2 | 5/5 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Light-activated AU-011) (N=3) | Cohort 2 (Single Medium Dose Light-activated AU-011) (N=3) | Cohort 3 (Single High Dose Light-activated AU-011) (N=3) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) (N=3) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) (N=3) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) (N=3) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) (N=3) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) (N=3) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) (N=12) | Cohort 10 (Observation Until Documented Growth of Tumor) (N=2) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) (N=5) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers) (N=13)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Light-activated AU-011) (N=3) | Cohort 2 (Single Medium Dose Light-activated AU-011) (N=3) | Cohort 3 (Single High Dose Light-activated AU-011) (N=3) | Cohort 4 (2 Repeat Medium Dose Light-activated AU-011) (N=3) | Cohort 5 (3 Repeat Medium Dose Light-activated AU-011) (N=3) | Cohort 6 (Single High Dose Light-activated AU-011 x 2 Lasers) (N=3) | Cohort 7 (3 Repeat High Dose Light-activated AU-011) (N=3) | Cohort 8 (3 Repeat High Dose Light-activated AU-011 x 2 Lasers) (N=3) | Cohort 9 (Expansion 3 Repeat High Dose Light-activated AU-011 x 2 Lasers) (N=12) | Cohort 10 (Observation Until Documented Growth of Tumor) (N=2) | Cohort 11 (2 Cycles of 3 Repeat High Dose Light-activated AU-011x2 Lasers) (N=5) | Cohort 12 (2 Cycles 3 Repeat High Dose Light-activatedAU-011x2lasers) (N=13)
Anterior chamber cell (Eye disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (5) | 1 (1) | 2 (3) | 2 (3)
Anterior chamber inflammation (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 3 (3) | 2 (4) | 8 (20) | 0 (0) | 4 (19) | 9 (19)
Conjuctival hemorrhage (Eye disorders) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (6) | 2 (3) | 6 (11) | 2 (2) | 5 (13) | 13 (26)
Conjuctival hyperemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (3) | 4 (4) | 2 (2)
Corneal edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Eye pain (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 3 | 5
Keratic precipitates (Eye disorders) | 1 | 2 | 1 | 2 | 1 | 0 (0) | 1 | 1 | 4 | 0 (0) | 1 | 2
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 1 | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 2 | 0 (0) | 2 | 0 (0) | 1 | 1
Ocular hypertension (Eye disorders) | 0 (0) | 1 | 1 | 0 (0) | 0 (0) | 1 | 0 (0) | 1 | 1 | 0 (0) | 0 (0) | 2
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 1 | 1 | 2 | 2 | 3 | 5
Retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 7 | 1 | 4 | 8
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 1 | 0 (0) | 0 (0) | 1
Visual acuity reduced (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 7 (11)
Vitreal cells (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 4 (4)
Vitreous floaters (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (5) | 1 (1)
Vitreous haze (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (8) | 1 (1) | 4 (6) | 0 (0) | 3 (5) | 4 (7)
Vitreous opacities (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Vitritis (Eye disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 3 (6) | 10 (16) | 1 (2) | 3 (11) | 9 (18)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (7)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Eyelid edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Iris adhesions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 2 (4) | 0 (0)
Retinal depigmentation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 2 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Intraocular pressured increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 1 (3) | 5 (9) | 8 (21)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 3 (7) | 1 (3)
Visual field defect (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSA states sites may publish or publicly disclose the results of the study after disclosure is given to the Sponsor for review at least 60 days prior to the date of submission for publication. Site agrees to discuss with Sponsor with respect to the presentation of study data and timing of the disclosure.

DOCUMENTS (2):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03052127/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03052127/SAP_001.pdf